CLINICAL TRIAL: NCT02350907
Title: Rapid Diagnosis of Antibiotic Resistance in Gonorrhoea: RaDAR-Go
Brief Title: Rapid Diagnosis of Antibiotic Resistance in Gonorrhoea
Acronym: RaDAR-Go
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 25/2013
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Gonorrhoea
Keywords: antimicrobial resistance; point-of-care testing; Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Swabs from the urethra, rectum, oropharynx, vagina and endocervix
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a laboratory-based assay that will be a real-time PCR test to detect the organism N. gonorrhoeae and its most important genetic markers of antimicrobial resistance. This study will also determine factors associated with gonorrhoea and describe sexual behaviours of men who have sex with men, to inform parameters for a mathematical model of gonorrhoea transmission and antimicrobial resistant gonorrhoea.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 years or above.
* Participant is literate in German, French, English or Hungarian.
* Participant is at risk for a N. gonorrhoeae infection. This is defined as:

  1. exhibiting signs/symptoms of a N. gonorrhoeae infection.
  2. having a sexual partner who has been diagnosed with a N. gonorrhoeae infection.
  3. participating in high-risk activities for a N. gonorrhoeae infection.

     Exclusion Criteria:
* Subject does not agree to undergo diagnostic test for gonorrhoea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and females at risk of gonorrhoea infection.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Presence of N. gonorrhoeae genetic markers for antimicrobial resistance in clinical specimens | Day of specimen sampling

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Low, Principal Investigator — University of Bern, Institute of Social and Preventive Medicine
Locations (3):
- Switzerland (3):
  - University Hospital of Bern, Bern
  - Ambulatorium Kanonengasse, Zurich
  - Checkpoint Zurich, Zurich

REFERENCES:
- [Background] Low N, Unemo M, Skov Jensen J, Breuer J, Stephenson JM. Molecular diagnostics for gonorrhoea: implications for antimicrobial resistance and the threat of untreatable gonorrhoea. PLoS Med. 2014 Feb 4;11(2):e1001598. doi: 10.1371/journal.pmed.1001598. eCollection 2014 Feb. PMID 24503544
- [Background] Fingerhuth SM, Bonhoeffer S, Low N, Althaus CL. Antibiotic-Resistant Neisseria gonorrhoeae Spread Faster with More Treatment, Not More Sexual Partners. PLoS Pathog. 2016 May 19;12(5):e1005611. doi: 10.1371/journal.ppat.1005611. eCollection 2016 May. PMID 27196299
- [Background] Dona V, Kasraian S, Lupo A, Guilarte YN, Hauser C, Furrer H, Unemo M, Low N, Endimiani A. Multiplex Real-Time PCR Assay with High-Resolution Melting Analysis for Characterization of Antimicrobial Resistance in Neisseria gonorrhoeae. J Clin Microbiol. 2016 Aug;54(8):2074-81. doi: 10.1128/JCM.03354-15. Epub 2016 May 25. PMID 27225407
- [Background] Low N, Unemo M. Molecular tests for the detection of antimicrobial resistant Neisseria gonorrhoeae: when, where, and how to use? Curr Opin Infect Dis. 2016 Feb;29(1):45-51. doi: 10.1097/QCO.0000000000000230. PMID 26658656
- [Result] Dona V, Smid JH, Kasraian S, Egli-Gany D, Dost F, Imeri F, Unemo M, Low N, Endimiani A. Mismatch Amplification Mutation Assay-Based Real-Time PCR for Rapid Detection of Neisseria gonorrhoeae and Antimicrobial Resistance Determinants in Clinical Specimens. J Clin Microbiol. 2018 Aug 27;56(9):e00365-18. doi: 10.1128/JCM.00365-18. Print 2018 Sep. PMID 29950339